CLINICAL TRIAL: NCT01957436
Title: A Prospective Randomised Phase III Study Of Androgen Deprivation Therapy With Or Without Docetaxel With Or Without Local Radiotherapy With Or Without Abiraterone Acetate And Prednisone In Patients With Metastatic Hormone-Naïve Prostate Cancer
Brief Title: A Phase III Study for Patients With Metastatic Hormone-naïve Prostate Cancer
Acronym: PEACE1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Janssen-Cilag Ltd. (Industry); European Organisation for Research and Treatment of Cancer - EORTC (Network); Ipsen (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0160/1105 GETUG AFU-21
Record Dates: First submitted 2013-09-24; First posted 2013-10-08 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Prostate Cancer
Keywords: prostate; cancer; metastatic hormone-naive; radiotherapy; abiraterone acetate; docetaxel
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Abiraterone Acetate; Radiotherapy; Androgen Antagonists; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A (Active Comparator): androgen deprivation therapy + docetaxel
  Interventions: Other: Androgen Deprivation Therapy; Drug: Docetaxel
- Arm B (Experimental): androgen deprivation therapy + docetaxel + abiraterone acetate + prednisone
  Interventions: Drug: abiraterone acetate; Other: Androgen Deprivation Therapy; Drug: Docetaxel
- Arm C (Experimental): Arm A + radiotherapy
  Interventions: Radiation: radiotherapy; Other: Androgen Deprivation Therapy; Drug: Docetaxel
- Arm D (Experimental): Arm B + radiotherapy
  Interventions: Drug: abiraterone acetate; Radiation: radiotherapy; Other: Androgen Deprivation Therapy; Drug: Docetaxel

INTERVENTIONS:
Drug: abiraterone acetate — abiraterone 1000mg/day (4 tablets of 250 mg (PO) per day) + prednisone 5mg bid
  Other Names: Zytiga
  Arms: Arm B; Arm D
Radiation: radiotherapy — 74 Gy in 37 fractions 3D-Conformal RT or Intensity Modulated RT (IMRT)
  Arms: Arm C; Arm D
Other: Androgen Deprivation Therapy — The ADT must consist in either LHRH agonist, LHRH antagonist or orchiectomy
Drug: Docetaxel — 6 cycles at 75mg/m²/cycle, one cycle every 3 weeks

SUMMARY:
This is a multi-center phase III study to compare the clinical benefit of androgen deprivation therapy with or without docetaxel with or without local radiotherapy with or without abiraterone acetate and prednisone in patient with metastatic hormone-naïve prostate cancer.

DETAILED DESCRIPTION:
Eligible patients can be randomize in the trial after his consent form has been signed, and after all inclusion and non-inclusion criteria have been checked.

The randomisation will result in the allocation of arm A (ADT +docetaxel), arm B (ADT +docetaxel +Abiraterone), arm C (ADT +docetaxel +radiotherapy) or arm D (ADT +docetaxel +Abiraterone +radiotherapy) in a 1:1:1:1 ratio.

The randomization will be stratified (by minimization) according to:

* enrolment center,
* performance status (0 vs. 1-2)
* disease extent: lymph nodes only vs. bone (with or without lymph nodes) vs. presence of visceral metastases.

CRPC is defined by cancer progression (either a confirmed PSA rise or a radiological progression) with serum testosterone being at castrated levels (<0.50 ng/mL).

When the CRPC stage is reached, castration (either LHRH agonist or LHRH antagonist) will be maintained in all patients.

Investigators will be free to manage patients reaching CRPC at their discretion (using for example docetaxel, zoledronic acid, denosumab, sipuleucel-T, radium-223, cabazitaxel, etc) according to local uses and guidelines.

Abiraterone may be used in arm A and C if abiraterone has become the standard treatment for CRPC when this stage is reached.

ELIGIBILITY:
Inclusion criteria:

1. Histologically or cytologically confirmed adenocarcinoma of the prostate,
2. Metastatic disease documented by a positive bone scan (any technique) or CT scan or an MRI. For patients with nodal metastases only, only patients with extra-pelvic enlarged lymph nodes (lymph nodes located above the iliac bifurcation) can be included if they have either:

   o At least one extra-pelvic lymph node ≥ 2 cm or extra-pelvic lymph node (s) ≥ 1 cm if the patients also have at least one pelvic lymph node ≥ 2 cm
3. Patients with ECOG ≤ 1 (patient with PS 2 due to bone pain can be accrued in the trial),
4. Life expectancy of at least 6 months,
5. Male aged ≥ 18 years old and ≤ 80 years old ,
6. Hematology values:

   * Hemoglobin ≥ 10.0 g/dL,
   * Platelet count ≥ 100,000/mL,
   * Neutrophil ≥ 1500 cells/mm³
7. Biochemistry values:

   * Renal function: Serum creatinine < 1.5 x ULN or a calculated creatinine clearance ≥ 60 mL/min,
   * Serum potassium ≥ 4 mmol/L,
   * Liver function:

     * Serum bilirubin ≤ 1.5 x ULN (except for patients with documented Gilbert's disease),
     * AST and ALT ≤ 1.5 x ULN (and ≤ 5 ULN in case of liver metastases),
   * ALK-P ≤ 2.5 x ULN (in case of bone metastasis, ALK-P<1000U/L if bilirubin is normal)
8. Patients must have received ADT for a maximum of 3 months before randomization and there must be a minimum of 6 weeks between the start of ADT and the start of Docetaxel,
9. Patients willing and clinically fit to receive Docetaxel which is defined by the following :

   * Patients respecting all inclusion and exclusion criteria And
   * Patients with no contraindication to docetaxel according to the SmPC of the drug And
   * Patients presenting all medical requirements to receive docetaxel according to the investigator's opinion.
10. Patients might have received previous radiation therapy directed to bone lesions,
11. Patients able to take oral medication,
12. Patients who have received the information sheet and signed the informed consent form,
13. Male patients who will receive Docetaxel and/or Abiraterone acetate and have partners of childbearing potential and/or pregnant partners must use a method of birth control in addition to an adequate barrier protection (condoms) as determined to be acceptable by the study doctor during the treatment period and for 4 weeks after the last dose of abiraterone acetate and/or for 6 months after the last dose of Docetaxel
14. Patients must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures,
15. Patients with a public or a private health insurance coverage, according to local laws for participation in clinical trials.

Exclusion Criteria:

1. Patients with previous definitive local treatment directed to the prostate primary cancer (radiotherapy, brachytherapy, radical prostatectomy, ultrasound, cryotherapy, or other). A previous trans-urethral resection of the prostate (TURP) and previous local treatments of metastases are allowed,
2. Prior cytotoxic chemotherapy or biological therapy for the treatment of prostate cancer,
3. Any chronic medical condition requiring a higher dose of corticosteroid than 5 mg prednisone/prednisolone twice daily,
4. Active infection or other medical condition for which prednisone/prednisolone (corticosteroid) use would be contra-indicated,
5. Previously treated with ketoconazole for prostate cancer for more than 7 days,
6. Prior systemic treatment with an azole drug (e.g. fluconazole, itraconazole) within 4 weeks of randomization,
7. Hypertension not controlled by an anti-hypertensive treatment (systolic BP ≥ 160 mmHg or diastolic BP ≥ 95 mmHg; 3 consecutive measures taken 5 minutes apart),
8. Severe or moderate hepatic impairment (Child - Pugh class C or B)
9. Active or symptomatic viral hepatitis or chronic liver disease (except Gilbert's disease),
10. History of pituitary or adrenal dysfunction,
11. Clinically known significant heart disease in the past 6 months as evidenced by myocardial infarction, or arterial thrombotic events, severe or unstable angina, or New York Heart association (NYHA) Class II-IV heart disease or cardiac ejection fraction measurement of < 50% at baseline,
12. Atrial Fibrillation, or other cardiac arrhythmia requiring therapy,
13. Patient with unstable pulmonary disease (eg. Pulmonary embolism)
14. Pathological finding consistent with small cell carcinoma of the prostate,
15. History of malignancy, except non-melanoma skin cancer, with a ≥ 30% probability of recurrence within 24 months,
16. Known allergies, hypersensitivity or intolerance to the study drugs or excipients or docetaxel
17. Administration of an investigational therapeutic within 30 days of randomization,
18. Patients already included in another therapeutic trial involving an experimental drug (patient in a non-experimental trial with no modification of the patient's care can be included),
19. Patients with significantly altered mental status prohibiting the understanding of the study or with psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule or any condition which, in the opinion of the investigator, would preclude participation in this trial. Those conditions should be discussed with the patient before registration in the trial,
20. Individual deprived of liberty or placed under the authority of a tutor.
21. Patients with impaired vision should undergo a prompt and complete ophthalmologic examination.

    Patients with Cystoid Macular Oedema cannot be included due to a potential risk of deterioration associated with docetaxel.
22. Concomitant use of strong CYP3A4 inhibitors (clarithromycin, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin.)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1173 (Actual)
Dates: Start 2013-11-13 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Survival | 7.5 years after the first inclusion
  Overall and radiographic progression-free survival in patients with metastatic hormone-naïve prostate cancer treated by androgen deprivation therapy and docetaxel
Survival | 9.5 years after the first inclusion
  Overall and radiographic progression-free survival in hormone-naïve prostate cancer patients with low metastatic burden whatever the standard of care received

SECONDARY OUTCOMES:
Castration resistance-free survival (CRFS) | 9.5 years after the first inclusion
Serious Genitourinary event-free survival (S-GU-EFS) | 9.5 years after the first inclusion
Prostate cancer specific survival | 9.5 years after the first inclusion
Time to next skeletal-related event | 9.5 years after the first inclusion
PSA response rate | 9.5 years after the first inclusion
Prospective correlative study of PSA response/progression at 8 months after initation of ADT | 9.5 years after the first inclusion
Time to pain progression | 9.5 years after the first inclusion
  will be evaluated by questionnaires
Time to chemotherapy for CRPC | 9.5 years after the first inclusion
Quality of life questionnaire - Core 30 (QLQ-C30) | At baseline, 6 months, 18 months, and at the end of treatment (up to 9.5 years)
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Functional Assessment of Cancer Therapy - Prostate (FACT-P) | At baseline, 6 months, 12 months, 18 months, and at the end of treatment (up to 9.5 years)
  The FACT-P is a self-assessment questionnaire to estimate the health-related quality of life in men with prostate cancer. This questionnaire, composed of 39 items consists of four subscales: Physical Well-Being (7 items), Social/Family Well-Being (7 items), Emotional Well-Being (6 items), Functional Well-Being (7 items), and prostate cancer subscale (12 items). Subscales are rated on 5-point Likert-type scale (from 0 = "Not at all" to 4 = "Very much"). For all subscales, a higher score represents better quality of life.
Toxicity (with a specific focus on the use of long-term low-dose steroids) | Throughout study completion, up to 9.5 years
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 4.0 (NCI-CTCAE v4.0) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.
Changes in bone mineral density | At baseline, 6 months, 12 months, and 24 months
  X-rays are used to measure how many grams of calcium and other bone minerals are packed into a segment of bone
Correlation of biomarkers with outcome | 9.5 years after the first inclusion
  Correlation of biomarkers with outcome, including the prognostic and predictive value on OS, rPFS and CRFS of a neuro-endocrine differentiation of the prostate cancer in the pathological specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Karim FIZAZI, Professor, Study Chair — Gustave Roussy, Cancer Campus Grand Paris - Paris; Alberto BOSSI, Doctor, Study Chair — Gustave Roussy, Cancer Campus Grand Paris - Paris
Locations (77):
- Belgium (6):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - Hôpitaux Universitaires Bordet Erasme- Institut Jules Bordet, Brussels
  - Hopital de Jolimont, Haine-Saint-Paul
  - AZ Groeninge Kortrijk - Campus Vercruysselaan, Kortrijk
  - Cliniques Universitaires Saint-Luc, Leuven
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
- France (49):
  - Clinique Claude Bernard, Albi
  - Institut de cancerologie de l'Ouest, Angers
  - Clinique Générale d'Annecy, Annecy
  - Institut Sainte Catherine, Avignon
  - Centre de la Baie, Avranches
  - Centre d'Oncologie et de Radiothérapie du Pays Basque, Bayonne
  - Chu Jean Minjoz, Besançon
  - Centre Pierre Curie, Beuvry
  - Institut Bergonie, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Hospitalier Alpes Leman, Contamine-sur-Arve
  - Chu de Mondor, Créteil
  - Centre Leonard de Vinci, Dechy
  - Centre Georges-François LECLERC, Dijon
  - Clinique Sainte Marguerite, Hyères
  - CHD Vendée, La Roche-sur-Yon
  - Clinique Victor Hugo, Le Mans
  - Chu de Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - CHU Lyon Sud, Lyon
  - Institut Paoli Calmettes, Marseille
  - Chu Timone, Marseille
  - Hôpital Nord, Marseille
  - Centre Azuréen de Cancérologie, Mougins
  - Centre Catherine de Sienne, Nantes
  - Centre Antoine Lacassagne, Nice
  - CHU Carémeau, Nîmes
  - CHR Orléans la source, Orléans
  - Institut Curie, Paris
  - Hôpital St Louis, Paris
  - Hopital TENON, Paris
  - Chic Quimper, Quimper
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Clinique Armoricaine de radiologie, Saint-Brieuc
  - CHU ST ETIENNE - Hôpital Nord, Saint-Etienne
  - CHP Saint Grégoire, Saint-Grégoire
  - Institut de Cancérologie del'Ouest - site René Gauducheau, Saint-Herblain
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - CENTRE DE CANCEROLOGIE Paris Nord, Sarcelles
  - Strasbourg Oncologie Libérale, Strasbourg
  - Hopitaux du Leman, Thonon-les-Bains
  - Centre Hospitalier Intercommunal de Toulon - La Seyne sur Mer - Hôpital Sainte Musse, Toulon
  - Institut Claudius Regaud, Toulouse
  - Clinique Pasteur, Toulouse
  - CHU de TOURS Hôpital Bretonneau, Tours
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Centre d'Oncologie Saint Yves, Vannes
  - INSTITUT GUSTAVE ROUSSY, Cancer Campus, Grand Paris, Villejuif
- Ireland (6):
  - Cork University Hospital, Cork
  - Adelaide and Meath incorporating National Children's hospital department, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - Mater Private Hospital, Dublin
  - St Vincent's University Hospital, Dublin
  - Galway University Hospital, Galway
- Italy (2):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - San Camillo Forlanini Hospitals, Roma
- Sc Radiotherapy Center Cluj SRL, Cluj-Napoca, Romania
- Spain (11):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital De la Santa Creu I Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Vall d'Hebron University Hospital, Barcelona
  - ICO Girona - Hospital Josep Trueta, Girona
  - Hospital Universitario HM Sanchinarro, Madrid
  - Althaia, Manresa
  - 'Hospital Clinico Virgen de la Victoria, Málaga
  - 'Parc Tauli Sabadell Hospital Universitari, Sabadell
  - Hospital Universitario de Salamanca, Salamanca
  - Institut Valenciano de Oncologia, Valencia
- Switzerland (2):
  - Fondation Dr. Henri Dubois-Ferrière Dinu Lipatti, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.

REFERENCES:
- [Derived] Alyamani N, Clementel E, Sargos P, Blanchard P, Supiot S, Ronchin P, Pommier P, Duberge T, Silva M, Hammoud Y, Hasbini A, Khalifa J, Gnep K, Scrase C, Saez J, Vieillevigne L, Christiaens M, Zilli T, Ribault H, Bossi A, Fizazi K, Andratschke N. Radiotherapy quality assurance for the PEACE 1 trial: An individual case review analysis. Radiother Oncol. 2025 May;206:110780. doi: 10.1016/j.radonc.2025.110780. Epub 2025 Feb 7. PMID 39924002
- [Derived] Roubaud G, Kostine M, McDermott RS, Bernard-Tessier A, Maldonado X, Silva M, Flechon A, Berthold DR, Ronchin P, Tombal BF, Mourey L, Gravis G, Escande A, Abadie-Lacourtoisie S, Maurina T, Climent MA, Ribault H, Bossi A, Foulon S, Fizazi K. Assessment of bone mineral density in men with de novo metastatic castration-sensitive prostate cancer treated with or without abiraterone acetate plus prednisone in the PEACE-1 phase 3 trial. Eur J Cancer. 2025 Mar 11;218:115293. doi: 10.1016/j.ejca.2025.115293. Epub 2025 Feb 6. PMID 39923274
- [Derived] Fizazi K, Foulon S, Carles J, Roubaud G, McDermott R, Flechon A, Tombal B, Supiot S, Berthold D, Ronchin P, Kacso G, Gravis G, Calabro F, Berdah JF, Hasbini A, Silva M, Thiery-Vuillemin A, Latorzeff I, Mourey L, Laguerre B, Abadie-Lacourtoisie S, Martin E, El Kouri C, Escande A, Rosello A, Magne N, Schlurmann F, Priou F, Chand-Fouche ME, Freixa SV, Jamaluddin M, Rieger I, Bossi A; PEACE-1 investigators. Abiraterone plus prednisone added to androgen deprivation therapy and docetaxel in de novo metastatic castration-sensitive prostate cancer (PEACE-1): a multicentre, open-label, randomised, phase 3 study with a 2 x 2 factorial design. Lancet. 2022 Apr 30;399(10336):1695-1707. doi: 10.1016/S0140-6736(22)00367-1. Epub 2022 Apr 8. PMID 35405085